CLINICAL TRIAL: NCT04470739
Title: Is Thymus Size of Infants Who Born to COVID-19 Positive Mothers Associated With Neonatal Morbidities?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seda Yilmaz Semerci, Neonatologist, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KSSEAH--CT
Record Dates: First submitted 2020-07-12; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Covid19; Thymic Hypoplasia
MeSH Terms: conditions — COVID-19; DiGeorge Syndrome | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infants born to COVID-19 positive mothers (Active Comparator): Infants, born to COVID-19 positive mothers, will be evaluated for cardiothymic index in their first chest X-ray.
  Interventions: Diagnostic Test: chest x-ray
- Infants born to COVID-19 negative mothers (No Intervention): Infants, born to COVID-19 negative mothers, will be evaluated for cardiothymic index in their first chest X-ray.

INTERVENTIONS:
Diagnostic Test: chest x-ray — First Chest X-ray in the first 6 hours of infants
  Arms: Infants born to COVID-19 positive mothers

SUMMARY:
COVID-19 infected pregnant women is thought to have variable degrees of inflammatory response against the disease. Investigators of present study, suggested that fetuses are affected from the possible fetal inflammatory syndrome in case of maternal COVID-19. Therefore the aim of his study is to evaluate that if the cardiothymic index is affected by the maternal COVID-19 and to demonstrate any possible association of this measurement with neonatal morbidities.

DETAILED DESCRIPTION:
COVID-19 infected pregnant women is thought to have variable degrees of inflammatory response against the disease. Fetus is known to be influenced by maternal systemic infections. Thymus size of fetus and the neonate, is proven to be changed by primarily inflammatory/infectious diseases. Investigators of present study, suggested that fetuses are affected from the possible fetal inflammatory syndrome in case of maternal COVID-19. Therefore the aim of his study is to evaluate that if the cardiothymic index is affected by the maternal COVID-19 and to demonstrate any possible association of this measurement with neonatal morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Infants born to COVID-19 positive or negative mothers
* Accepted to participate with an informed consent
* Infants who required to get chest X-ray within the first 6 hours

Exclusion Criteria:

* Infants whose mothers' have any kind of acute or chronic systemic disease or inflammation/infection
* Lack of an informed consent
* Infants who did not require to get chest X-ray within the first 6 hours

Max Age: 7 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2020-05-30 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Cardiothymic index | 4 months
  Cardiothymic index will be measured by using the thymic shadow divided by largest diameter of mediastinum in the chest X-ray of those infants.

SECONDARY OUTCOMES:
Immune profile | 6 months
  In long term follow up of those patients, infants will be evaluated for any kind of immune deficiency or quantitative or qualitative abnormalities of leukocytes

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No